CLINICAL TRIAL: NCT02977689
Title: Phase 2 Study of IDH305 in Subjects With IDH1 Mutant Grade II or III Glioma That Has Progressed After Observation or Radiation Therapy
Brief Title: Trial of IDH305 in IDH1 Mutant Grade II or III Glioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis paused all study start-up activities due to safety evaluation of IDH305 compound.
Sponsor: NYU Langone Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-00589
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Glioma
Keywords: Isocitrate dehydrogenase (IDH); R-2-Hydroxyglutarate (2-HG); Gene encoding UDP-glucuronosyltransferase (UGT1A1); Glioblastoma (GBM); IDH305; IDHR132 mutations; Astrocytoma; Oligodendroglioma; Oligoastrocytoma; IDH1 R132H; IDH1
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IDH305 (Experimental): IDH305 550 mg, oral, two times per day
  Interventions: Drug: IDH305

INTERVENTIONS:
Drug: IDH305 — study drug used to inhibit IDH1 mutation in these tumors, resulting in anti-tumor activity.

SUMMARY:
The purpose of this study is to found out if the drug IDH305 is safe and effective in subjects with IDH1 mutant grade II or III glioma that has progressed after observation or radiation therapy.

DETAILED DESCRIPTION:
IDH305 is an orally available, brain-penetrant, mutant-selective allosteric IDH1 inhibitor that blocks mutant IDH1-dependent production of 2-HG.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements.
2. Subject must be ≥18 years of age.
3. Patients must have written documentation of IDH1 mutation at the R132 locus by immunohistochemistry or DNA sequencing in their tumor.
4. Histopathological diagnosis of a glioma of WHO grade II or III at initial diagnosis. Documentation of diagnosis by pathology report is sufficient for eligibility.
5. First line management with observation alone or external beam radiation after surgery. Notes or records from the treating oncologist or radiation oncologist are required for documentation of treatment history.
6. Patients must have unequivocal progression on brain MRI after observation or external beam radiation. If a patient was initially diagnosed with a non-enhancing tumor and the tumor develops new contrast-enhancement at progression, they will be excluded except for the following exceptions:

   1. Patients with tumors that were contrast-enhancing at initial diagnosis of grade II or III glioma will be allowed if their tumors are contrast-enhancing at progression as well.
   2. If a patient with a grade II or III glioma has a tumor that develops new contrast-enhancement at progression, the enhancing portion of the progressive tumor must be biopsy proven WHO grade II or III at progression.
7. Measurable tumor of at least 1 cm x 1 cm in diameter by MRI. The measurable tumor may be contrast-enhancing or non-enhancing.
8. Interval of at least 12 weeks from the completion of any prior radiotherapy and registration. If patients have not passed an interval of at least 12 weeks, they may still be eligible if they meet one or more of the following criteria:

   1. New areas of tumor outside the original radiotherapy fields as determined by the investigator, or
   2. Histologic confirmation of tumor (as opposed to pseudo-progression or radiation necrosis) through biopsy or resection
9. Collection of an archival tumor block with a minimum of 1 cm2 surface area of viable tumor or at least 20 unstained 5 micron slides from the most recent surgery.
10. Karnofsky performance status (KPS) ≥60.
11. An interval of at least 2 weeks (to start of study agent) between prior surgical resection of glioma, or one week for stereotactic biopsy of glioma.
12. Adequate hematologic, hepatic, and renal function defined by absolute neutrophil count ≥1.0 x 109/L, hemoglobin ≥8 g/dL, platelet count ≥ 75 x 109/L (may have been transfused), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN), total bilirubin > 1 x ULN, and serum creatinine >1.5 x ULN

Exclusion Criteria:

1. Glioblastoma (WHO grade IV) histopathology on any tumor sample
2. Leptomeningeal gliomatosis
3. Unable to tolerate a contrast-enhanced brain MRI or if MRI is contraindicated
4. Two weeks since any major surgery treatment (mediastinoscopy, insertion of a central venous access device and insertion of a feeding tube are not considered major surgery) prior to registration, with the exception of stereotactic biopsy for glioma, in which case an interval of 1 week until registration is allowed.
5. Patients who are currently receiving treatment with a prohibited medication or herbal remedy that cannot be discontinued at least one week prior to the start of treatment.

   1. Narrow therapeutic index substrates of CYP3A, CYP2C9, CYP2C19, and CYP2C8
   2. Medications, herbs and supplements that are strong inhibitors and strong inducers of CYP3A
   3. Other herbal preparations and supplements
   4. Inhibitors of UGT1A1
6. Prior exposure to a therapy targeting IDH1, including targeted inhibitors of IDH1 and anti-IDH1 vaccines.
7. Prior treatment with any cytotoxic chemotherapy, including but not limited to temozolomide, lomustine, Nimustine Hydrochloride (ACNU), bis(chloroethyl) nitrosourea (BCNU), procarbazine, vincristine, carboplatin, irinotecan, Gliadel wafer, cyclophosphamide, etoposide, etc. Chemotherapy is associated with hypermutation phenotype at recurrence and therefore patients who have had prior treatment with these agents are excluded.
8. Rapidly progressing neurological symptoms related to underlying disease requiring increasing doses of corticosteroids. Steroid use for management of gliomas is allowed but the dose must be stable for at least 1 week preceding the baseline MRI/CT. If the corticosteroid dose is increased between the date of imaging and the initiation of study treatment, a new baseline MRI is required.
9. Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within the prior 2 years from the time of registration; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
10. Patients with corrected QT using the Fridericia correction (QTcF) > 470 msec, or other clinically significant, uncontrolled heart disease, including acute myocardial infarction or unstable angina < 3 months prior to the first dose of IDH305.
11. Any other medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures such as the presence of other clinically significant cardiac, respiratory, gastrointestinal, renal, hepatic, infectious, psychiatric or neurological disease.
12. Patients with Gilbert's syndrome or other heritable diseases of bile processing.
13. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
14. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 30 days after the use of the investigational medication. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that patient
    * Combination of any two of the following (a+b, a+c, or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal, for example hormone vaginal ring or transdermal hormone contraception.

         * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
15. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
16. Sexually active males must use a condom during intercourse while taking the drug and for 30 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via semen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Radiographic response rate | up to 8 weeks

SECONDARY OUTCOMES:
Safety (adverse events) of the protocol therapy | up to 2 years
  The adverse events are evaluated per Common Terminology Criteria for Adverse Events (CTCAE) 4.03
Volumetric radiographic response rate | up to 6 months
Median duration of response | up to 6 months
Median progression-free survival (PFS) | up to 6 months
Progression-free survival at 6 months (PFS6) | up to 6 months
2-year overall survival (OS) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Chi, MD, PhD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- Laura & Isaac Perlmutter Cancer Center & NYU Langone Medical Center, New York, New York, United States